CLINICAL TRIAL: NCT05943834
Title: Early Detection of Alzheimer's Disease and Affective Disorders by Automated Voice and Speech Analysis
Brief Title: Early Detection of Alzheimer's Disease and Affective Disorders by Automated Voice and Speech Analysis (PLATA)
Acronym: PLATA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23-PP-03
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurocognitive Disorders
Keywords: Alzheimer's disease; Mood disorder
MeSH Terms: conditions — Neurocognitive Disorders; Alzheimer Disease; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a minor or major neurocognitive disorder: Every patient will receive one semi-automated phone call, during the call a series of cognitive tasks will be performed.
  Each task will be recorded in a secondary audio stream which records the participant responses to allow for deep speech analysis of performance on these tasks
  Interventions: Other: Series of cognitive tasks during a semi-automated call

INTERVENTIONS:
Other: Series of cognitive tasks during a semi-automated call — Tasks:
  * Verbal learning recall (immediate) or Story Recall task (immediate)
  * Narrative Storytelling /free speech
  * Verbal fluency task
  * Verbal learning recall (delayed) or Story Recall task (delayed)

SUMMARY:
PLATA aims to develop an algorithm to identify vocal biomarkers of Alzheimer's dementia.

Using data collected as part of routine care, speech patterns will be compared to known biomarkers of Alzheimer's disease, such as amyloid 1-42 and p-Tau in CSF (cerebrospinal fluid).

If biomarkers of speech can be identified in Alzheimer's disease, it is possible that patients and research participants will no longer need to undergo need to undergo the intensive and invasive baseline biomarker methods currently used, such as lumbar punctures and PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Diagnosis relevant biomarker and neuropsychological data already available
* Cognitively healthy to very mild dementia (CDR score max. 0.5)
* Sufficient knowledge of the study language to understand study information, non opposition form,and questionnaires
* Expression of non opposition

Exclusion Criteria:

* Hearing problems
* Patient protected by law, under guardianship or curator ship, or not able to participate in a clinical study according to the article L.1121-16 of the French Public Health Code

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through the Memory Clinic at the Geriatric Hospital in Nice (Centre de Mémoire de Ressources et de Recherche, CHU de Nice, Institut Claude Pompidou 10 rue Molière, 06 100 NICE) with a minor or major neurocognitive disorder whose etiology is either:
  * Probable Alzheimer's disease (positive AD biomarkers)
  * Mood disorder
  * Not related to a mood disorder and with negative AD biomarkers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Build and validate speech-based machine learning models for relevant Phenotype detection through access to phenotyped patients from reference memory center. | 20 minutes
  Speech biomarker algorithm(s)

CONTACTS AND LOCATIONS:
Overall Officials: Eric ETTORE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No